CLINICAL TRIAL: NCT00807287
Title: Evaluation of Two Methods of Jejunal Placement of Enteral Feeding Tubes in Critically Ill Patients: Endoscopic Versus Unguided, Frictional Method
Brief Title: Evaluation of Two Methods of Jejunal Placement of Enteral Feeding Tubes in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Ulrike Holzinger, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 517/2004
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Critically Ill
Keywords: jejunal tube placement
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Placement of jejunal feeding tube using the unguided frictional method
  Interventions: Procedure: Jejunal tube placement using the unguided frictional method
- 2 (Active Comparator): Jejunal tube placement using the endoscopic method
  Interventions: Procedure: Jejunal tube placement using the endoscopic method

INTERVENTIONS:
Procedure: Jejunal tube placement using the unguided frictional method — The self-advancing nasal jejunal feeding tube has small alternating cilia-like plastic flaps to help to advance it into the small bowel via peristalsis. The tube is placed in the stomach (50-60 cm mark). Then the tube is left in place for 1 hour to allow the patient's peristalsis to advance the tube by catching its small plastic tabs. Thereafter, the tube is manually advanced 10 cm every hour until the 100 cm mark of length is reached. To improve peristalsis, 10mg metoclopramide i.v. and 200mg erythromycin i.v. 15 minutes before the procedure are administered.
  Other Names: Tiger Tube TM (Cook® Medical Inc., Bloomington, USA)
  Arms: 1
Procedure: Jejunal tube placement using the endoscopic method — Jejunal feeding tubes are placed using endoscopy
  Other Names: Freka® Trelumina (Fresenius Kabi AG, Bad Homburg, Germany)
  Arms: 2

SUMMARY:
In patients with high gastric residual volumes jejunal feeding is recommended. Jejunal feeding tubes can be placed in different ways. The endoscopic technique yields a success rate between 90 and 98% for a correct jejunal placement. However, it requires endoscopic equipment and trained staff. In contrast in small uncontrolled trials different unguided techniques resulted in success rates up to 75%, only. In this prospective randomized trial the success rate of a correct jejunal placement with the endoscopic technique is compared with the unguided frictional technique. The investigators hypothesize that the success rate of the unguided frictional placement method will be lower than the success rate of the endoscopic method.

DETAILED DESCRIPTION:
Artificial nutrition is an important link between the response to injury and recovery in critically ill patients admitted to an intensive care unit (ICU) Therefore artificial nutrition has become a part of ICU standard-therapy.

Enteral nutrition (EN) has shown to be superior to total parenteral nutrition. Consequently, EN should be first choice in patients without contraindications for enteral feeding. However, although EN is beneficial for the patient it may also be associated with complications because of gastroduodenal motility disorders, which are common in critically ill patients, especially when they receive analgosedation.

Clinical studies have shown that up to 62,8% of patients receiving EN have gastrointestinal complications like high gastric residuals (≥200ml), vomiting, abdominal distension and regurgitation. These complications lead to interruptions of the EN, which result in a low caloric intake of the patient.

In order to avoid at least some of these complications the American Society of Chest Physicians consensus statement recommends small bowel feeding if gastric residual volumes of 150ml or higher occur. The Canadian clinical practice guidelines recommend acceptance of gastric residual volumes up to 250 ml, use of prokinetic agents and jejunal feeding for patient, who are at high risk for intolerance of EN (on inotropes, sedatives, paralytic agents.

Small bowel feeding is the best method to feed the patient enterally because it is associated with a significant decrease of reflux, a reduced risk of aspiration and an adequate caloric intake.

For small bowel feeding the placement of a jejunal feeding tube is necessary. There are several possibilities to place the tube in the small bowel. An excellent method is endoscopy, which has a success rate up to 98% and moreover allows an evaluation of the upper GI-tract concerning pathologies. However it is a rather time consuming procedure, which is of limited availability and requires trained staff. As more simple alternatives unguided tubes, which place themselves in the small bowel were tested and showed success rates up to 75% only. Different patient population and different severity of illness in ICU patients mislead to this developed difference in success rate.

So far a prospective randomised trial comparing the endoscopic method versus the unguided frictional placement has not been studied. Therefore the aim of the study is the evaluation of the success rate of jejunal placement of these two different methods in a comparative ICU patient population. The secondary outcome parameters are: time to successful placement, time in place, costs and complications. We hypothesize that the success rate of the unguided frictional placement method will be lower than the success rate of the endoscopic method.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanically ventilated
* Intolerance of intragastric enteral nutrition: defined as high gastric residual volumes (≥ 250ml / 24 hours) and/or repeated vomiting.

Exclusion:

* Contraindication for enteral nutrition or gastric endoscopy
* Previous upper gastrointestinal surgery
* Signs of active gastric bleeding
* Severe nasopharyngeal injuries or stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-02; Primary Completion 2006-02 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Success rate of correct jejunal placement | 24h

SECONDARY OUTCOMES:
Duration of jejunal tube placement (initiation of jejunal tube placement till correct jejunal placement | 24h
Adverse effects of tube placement and adverse side effects of jejunal tubes during the ICU stay | ICU-stay

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Holzinger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria